CLINICAL TRIAL: NCT02951403
Title: Results of the Treatment of Patients With Elbow Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Central Finland Hospital District (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R15117
Record Dates: First submitted 2016-06-06; First posted 2016-11-01 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Elbow Osteoarthritis
Keywords: elbow arthroscopy; DASH; elbow locking; elbow osteoarthritis
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative treatment (Experimental): Patients to whom the elbow arthroscopy will be performed.
  Interventions: Procedure: Elbow arthroscopy
- Conservative treatment (Other): Patients to whom special physiotherapy will be advised.
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Procedure: Elbow arthroscopy — Arthroscopic debridement, osteophyte excision, loose body extirpation is carried on to patients.
  Arms: Operative treatment
Other: Conservative treatment — Physiotherapy protocol is introduced to patients.
  Arms: Conservative treatment

SUMMARY:
The study is a prospective case controlled clinical trial. The purpose of the study is to investigate the effect of elbow arthroscopy in the treatment for osteoarthritis of the elbow when compared to conservative treatment.

DETAILED DESCRIPTION:
Patients will be recruited at departments of hand surgery and orthopedic surgery outpatient clinics. The control group will be patients to whom the conservative treatment continues. Patients who meet the inclusion criteria will be asked to participate and sign the informed consent. Therefore the investigators have two treatment groups: group 1 who receives an elbow joint debridement arthroscopically without physiotherapy and group 2 who receives only conservative treatment with physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic post-traumatic or primary osteoarthritis - mechanical locking and/or decreased range of motion ( >30°)
* Radiographic evidence of at least mild primary or post-traumatic osteoarthritis according to Broberg - Morrey classification symptoms lasting at least 6 months
* Patients willingness to participate the study
* All patients 18-80 ages

Exclusion Criteria:

* Patients with previous severe soft tissue trauma at elbow region ( crush, burns etc - the elbow joint problems are not joint specific)
* Patients with crystal arthropathy or inflammatory arthritis
* Patient refuses to participate the study
* Patients with dementia or are institutionalized
* Patients with severe substance addiction
* Patient does not understand written and spoken guidance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Quick DASH score | 24 Months

SECONDARY OUTCOMES:
VAS score | 24 Months
Range of motion | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ville Mattila, MD, PhD, Study Chair — professor; Margit Karelson, MD, Principal Investigator — hand surgeon
Locations (3):
- Finland (3):
  - Central Finland Central Hospital, Jyväskylä
  - Tampere University Hospital, Tampere
  - Tampere University Hospital, Hatanpää, Tampere

IPD SHARING:
Plan to Share IPD: No